CLINICAL TRIAL: NCT06318650
Title: Evaluation of Post Extraction Hard Tissue Alteration Following Ridge Preservation in the Esthetic Zone Using Allogeneic Dentin Matrix Versus Demineralized Freeze-Dried Bone Allograft: A Randomized Controlled Clinical Trial
Brief Title: Post Extraction Changes After Ridge Preservation Using Allogeneic Dentin Matrix Vs Demineralized Freeze Dried Allograft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatima Mubarak Saleem Bin Nuhaid, Principal Investigator Fatima Mubarak Master Degree student, Periodontology department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19124PER6_3_1
Record Dates: First submitted 2024-03-11; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Socket Preservation
Keywords: Socket preservation; Ridge preservation; Allogeneic dentin matrix; Demineralized freeze dried bone allograft; DFDBA
MeSH Terms: interventions — Demineralized Dentin Matrix

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogenic Demineralized Dentin Matrix (Experimental): Following atraumatic tooth extraction, curettes will be used to remove granulation tissues, and the socket will be irrigated with sterile normal saline.Then the socket will be filled with Allogeneic Dentin Matrix (that has been prepared before) to the crestal level of then bone followed by placement of a collagen membrane to cover the socket. Suturing technique will be a criss-cross horizontal mattress to ensure that most of the grafting material is covered.
  Interventions: Biological: Demineralized Dentin Matrix
- Demineralized Freeze-Dried Bone Allograft (Active Comparator): Following atraumatic tooth extraction, curettes will be used to remove granulation tissues, and the socket will be irrigated with sterile normal saline.Then the socket will be filled with Demineralized freeze-dried bone allograft (DFDBA) to the crestal level of then bone followed by placement of a collagen membrane to cover the socket. Suturing technique will be a criss-cross horizontal mattress to ensure that most of the grafting material is covered.
  Interventions: Biological: Demineralized freeze-dried bone allograft (DFDBA)

INTERVENTIONS:
Biological: Demineralized Dentin Matrix — preparation of Allogenic Demineralized Dentin Matrix: Extracted teeth will be collected from the Departments of oral maxillofacial surgery and periodontics, Cairo university. Cleaning the teeth from any caries, Filings, cement, tartar, soft tissue debris and prosthetic components will be performed using a diamond bur under abundant irrigation with physiological water. Then it will be proceeded to the following steps
  1. (Washing with Distilled water ) 2. (Quick Freezing with liquid nitrogen, then Grinding to particle size of 300- 800 μm). 3.(Ultrasonic Cleaning cycles, 1st with Distilled water , 2nd with 5-7% Hydrogen Perioxide then 3rd with Distilled water for at 60-80 o) 4. (Defatting with Chloroform Methanol Solution1:0.5. 5. (Demineralization with0.5N HCL) 6. (Dehydration with Neutral Ethyl Alcohol then Defatting with Chloroform Methanol Solution 1:0.5 for ) 7. (Washing with Normal Saline & Freeze Drying then Sterilization using Ethylene oxide gas).
  Arms: Allogenic Demineralized Dentin Matrix
Biological: Demineralized freeze-dried bone allograft (DFDBA) — combination allograft, is a particulate bone graft combining 70% mineralized ground cortical with 30% demineralized ground cortical Particle sizing: 250 - 1000um.
  Arms: Demineralized Freeze-Dried Bone Allograft

SUMMARY:
the aim of this study is to establish if there are clinical, radio-graphical and histomorphometrical differences between using Allogenic Demineralized Dentin matrix versus Demineralized Freeze-Dried Bone Allograft (DFDBA) as a clinical application in alveolar bone regeneration procedures related to implant dentistry, including socket preservation, alveolar ridge augmentation, after tooth extraction in the esthetic zone.Will ridge preservation using Allogeneic Dentin Matrix be more effective than Demineralized Freeze-Dried Bone Allograft in managing the post extraction hard tissue alterations?

The initial therapy consists of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques. alginate impression will be taken to fabricate an acrylic stent to be used as reference for measurements of width of ridge clinically.

Flapless and atraumatic tooth extraction will be initiated, Then the socket will be filled either with Allogeneic Dentin Matrix or Demineralized freeze-dried bone allograft (DFDBA) up to the crestal level of then bone followed by placement of a collagen membrane to cover the socket. criss-cross horizontal mattress suturing technique

Intervention group: The socket will be filled with Allogeneic Dentin Matrix Control group: The socket will be filled with Demineralized freeze-dried bone allograft (DFDBA).

For both groups, All the subjects will be evaluated at pre-surgical, baseline and 6 months post surgical months for clinical parameters and baseline( immediate post-surgical and 6 months post-surgical . Outcomes: Change in ridge width clinically after 6 months, Change in the radiographic buccal vertical bone level, Change in the radiographic palatal vertical bone level,Change in the radiographic horizontal bone level,Percentage of new vital bone formation,Percentage of residual bone graft and Implant Primary Stability.

DETAILED DESCRIPTION:
This study aims to evaluate clinical, radiographic and histomorphometrical differences between using Allogenic Demineralized Dentin matrix versus Demineralized Freeze-Dried Bone Allograft (DFDBA) in alveolar ridge preservation after tooth extraction in the esthetic zone.

Research Procedure in brief:

The study is to be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry- Cairo University, Egypt.Patients are to be selected from the outpatient clinic of the department of Oral Medicine and Periodontology, clinic of the department of Oral surgery and clinic of the department of Endodontics -Cairo University.

The initial therapy consists of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques.

surgical interventions: Atraumatic extraction.The patient will rinse their mouth with 0.12% Chlorhexidine Administration of 4% articaine hydrochloride with 1:100,000 epinephrine will be as local anesthetic agent.Flapless and atraumatic tooth extraction will be initiated, using 15C blade intrasulcular incision will be performed.A periotome will be utilized to sever the periodontal ligament (PDL) fibers, followed by extraction witha straight elevator and extraction forceps.

Test group:

preparation of Allogenic Demineralized Dentin Matrix. Extracted teeth will be collected from the Departments of oral maxillofacial surgery and periodontics, Cairo university. Cleaning the teeth from any caries, Filings, cement, tartar, soft tissue debris and prosthetic components will be performed using a diamond bur under abundant irrigation with physiological water. Then it will be proceeded to the following steps

1. (Washing with Distilled water for 30-120 mins) The dental root that has had its soft and pulp tissues removed is cleaned with distilled water for anywhere between 30 minutes and two hours. The dental root includes residual dentin and cementum, even though soft and pulp tissues have been removed.
2. (Quick Freezing with liquid nitrogen -160 o C for 30-120 mins Then Grinding to particle size of 300- 800 μm) The dental root is processed into powder by quick-freezing and crushing, the same method used for the dental crown, with an average particle diameter of 200 mm to 1,500 mm. To eliminate impurities and remaining soft tissue, the powder will be washed with distilled water for 30 minutes to 2 hours.
3. (Ultrasonic Cleaning cycles, 1st with Distilled water for 5-10 mins, 2nd with 5-7% Hydrogen Perioxide10-30 mins then 3rd with Distilled water for 5-10 mins at 60-80 o) Each cycle of ultrasonic cleaning includes: a first washing step in which the powder is processed with ultrasonic cleaning for about 5 minutes to about 10 minutes in pure water or sterilized distilled water; a second washing step in which the powder is processed with ultrasonic cleaning for about 10 minutes to about 30 minutes in hydrogen peroxide solution; and a third washing step in which the powder is processed with ultrasonic cleaning for about 10 minutes to about 30 minutes in hydrogen peroxide solution. The concentration of the hydrogen peroxide solution is around 5% to 7%, the volume of the washing fluid of each washing step is approximately 5 times to approximately 10 times that of the powder, and the temperature of the washing fluid may be approximately 60°C to 80°C.
4. (Defatting with Chloroform Methanol Solution1:0.5 for 3-12 hours) The powder cleaned in the preceding step can be largely degreased using a chloroform methanol solution with a chloroform to methanol weight ratio of about 1:0.5 to about 1:2 for 3 to 12 hours. The largely degreased powder can be centrifuged to remove floating fat and rinsed with distilled water for at least 1 hour.
5. (Demineralization with0.5N HCL for 10-60 mins) For about 10 minutes to about 1 hour, the principally degreased powder is delimed (Demineralized) with about 0.5N hydrochloric acid aqueous solution whose volume is about 5 times to about 10 times that of the powder.
6. (Dehydration with Neutral Ethyl Alcohol for 30 mins then Defatting with Chloroform Methanol Solution 1:0.5 for 3-12 hours) The delimed powder is next dehydrated with neutral ethyl alcohol for 30 minutes to 2 hours. The dehydrated powder can be secondary degreased using a chloroform methanol solution with a chloroform to methanol weight ratio of approximately 1:0.5 to about 1:2 for 3 to 12 hours.
7. (Washing with Normal Saline & Freeze Drying then Sterilization using Ethylene oxide gas) The above-mentioned powder is degreased, delimed, and dehydrated before being post-treated with the steps of washing with normal saline solution and freeze-drying the degreased, delimed, and dehydrated powder; and sterilization will be done using ethylene oxide gas.

Alveolar ridge preservation:

* Following extraction, curettes will be used to remove granulation tissues, and the socket will be irrigated with sterile normal saline.
* Then the socket will be filled either with Allogeneic Dentin Matrix or Demineralized freeze-dried bone allograft (DFDBA) in control group up to the crestal level of then bone followed by placement of a collagen membrane to cover the socket. Suturing technique will be a criss-cross horizontal mattress to ensure that most of the grafting material is covered.

Postoperative Care and follow up:

* Participants will be instructed to avoid causing any damage to the operated site, to prevent interfering with the sutures, and to avoid consuming hot meals or vigorous rinsing.
* They will be encouraged to continue cleaning their teeth, only avoiding the operated site. Moderate tooth brushing for the operation site will be recommended after two weeks.
* Participants will be given Amoxicillin 500 mg three times a day for seven days, or doxycycline 100 mg twice a day if they are penicillin sensitive.
* Ibuprofen 600 mg will be provided for severe pain.
* Participants will be asked to use a 0.12% Chlorhexidine mouthwash twice daily for two weeks to assist gentle rinsing.
* Sutures will be removed two weeks after the surgery.
* A baseline cone-beam computed tomography (CBCT) scan will be conducted on the same day postoperative. A final follow-up visits and CBCT scan will be scheduled for six months postoperative to evaluate the dimensions of the alveolus before implant placement.

Biopsy collection After a 6-months healing period, a biopsy will be collected from the central area of the grafted site with a 3- mm trephine bur at the time of implant implantation. The biopsy will be immediately fixed in 10% neutral buffered formalin, followed by dehydration in a series of increasing concentration alcohol baths (varying from 50% to 100%). The specimen will then be encased in paraffin. Finally, a 4 m thick tissue section will be cut and stained with hematoxylin and eosin for subsequent histological investigation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the age of 20-55.
* Single rooted, non-restorable or hopeless tooth with adjacent teeth.
* Extraction socket with no more than 50% buccal bone loss
* Patients accept 6-months follow-up period (cooperative patients).
* Patients provide an informed consent.

Exclusion Criteria:

* Patients with uncontrolled systemic disease.
* Patient with severe para-functional habits.
* Patients with poor maintenance of oral hygiene.
* Pregnancy.
* Smokers.
* Patients taking any medications that could compromise healing.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Ridge width over 6 months | after 6 months postoperatively
  Before surgical intervention, baseline and 6-month postoperative examination will be conducted. Before surgical procedure ridge width will be measured using caliper, a resin acrylic stent will be placed measurements of 3mm and 5mm from gingival margin will be marked and measures the ridge width through it, this will be repeated after extraction (baseline) and 6 months postoperative.

SECONDARY OUTCOMES:
Change in the radiographic vertical bone level | after 6 months postoperatively
  Baseline and 6-month postoperative CBCT scans will be conducted. At both time points, measurements will be taken with identical reference points and lines. The most apical point of the extraction socket will be determined on the baseline image, and two reference lines will be created to form a reference. The vertical reference line will cross the apical reference point at the midway of the extraction socket.The alveolus' height will be measured at the midbuccal aspect (BH) and the midlingual aspect (LH).
Change in the radiographic horizontal bone level | after 6 months postoperatively
  CBCT scans will be performed at baseline and 6 months thereafter. At both time points, measurements will be taken with identical reference points and lines. The most apical point of the extraction socket will be determined on the baseline image, and two reference lines will be created to form a reference. The vertical reference line will cross the apical reference point at the midway of the extraction socket. In addition, a horizontal reference line perpendicular to the vertical line will be drawn, passing through the apical reference point.The horizontal ridge width will be measured at three different levels: 1 mm, 3 mm, and 5 mm below the crest's most coronal aspect. These measurements will be denoted by the letters HW-1, HW-3, and HW-5.
Percentage of new vital bone formation and residual graft | after 6 months postoperatively
  The biopsies will be preserved in a 10% formalin solution. Following that, they will undergo four weeks of EDTA decalcification. The specimens will be treated and embedded in paraffin after decalcification to generate tissue blocks. The paraffin blocks will be split into longitudinal sections of 5m thickness. For histological examination and histomorphometric analysis, these slices will be stained with hematoxylin and eosin (H&E) or Masson's trichromatic (MT) stains. A digital light microscope will be used to photograph the stained sections.
Implant Primary Stability | after 6 months postoperatively
  The Osstell Mentor Resonance Frequency Analyzer (Osstell AB, Goteborg, Sweden) will be used to evaluate the primary stability of the implant fixture. For each implant, two measurements will be collected in the buccolingual and mesiodistal directions. The representative implant stability quotient (ISQ) for each particular implant will be calculated as the average of these two measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Manal M. Hosny, Professor, Study Director — Cairo University; Fatima M. Saleem Bin Nuhaid, Bachelor, Principal Investigator — Cairo University; Weam A. El-Battawy Study Chair, Ass. Prof., Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt